CLINICAL TRIAL: NCT06134661
Title: Optimizing rTMS for Psychomotor Slowing in Psychosis (ATMSSlowing) - A 1-week, Non-randomised Clinical Trial of add-on Accelerated Repetitive Transcranial Magnetic Stimulation for Psychomotor Slowing in Psychosis
Brief Title: Accelerated rTMS for Psychomotor Slowing
Acronym: ATMSSlowing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Planned interim analyses demonstrated that the main aim of the study was already met. Recruitment was stopped. Early termination was unrelated to safety.
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATMSSlowing
Record Dates: First submitted 2023-10-23; First posted 2023-11-18 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Schizophrenia; Psychosis; Schizophrenia and Related Disorders; Schizo Affective Disorder; Brief Psychotic Disorder
Keywords: Psychomotor Slowing
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Psychomotor Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm: Treatment with cTBS (Experimental): This is a single-arm study. All participants will receive the treatment with cTBS.
  Interventions: Device: cTBS (continuous Theta Burst Stimulation)

INTERVENTIONS:
Device: cTBS (continuous Theta Burst Stimulation) — Continuous Theta Burst Stimulation (cTBS) is an inhibitory stimulation protocol of the Transcranial Magnetic Stimulation (TMS) device that temporarily inhibits brain activation in a small targeted brain area.
  The investigators apply the cTBS protocol 3 times daily at 100% of the resting motor threshold (RMT) for 1500 pulses per session.
  Other Names: TMS (Transcranial Magnetic Stimulation)

SUMMARY:
The goal of this clinical trial is to optimize the treatment of psychomotor slowing in patients with schizophrenia using Transcranial Magnetic Stimulation (TMS). A previous randomized controlled trial indicated that inhibitory stimulation over the supplementary motor area (SMA) once daily over 3 weeks ameliorates psychomotor slowing. In this trial the investigators use a shorter inhibitory protocol called cTBS and to be applied 3 times per day. This should lead to faster treatment response and less burden to patients.

The main question the investigators aim to answer are:

Can the treatment with cTBS 3 times per day ameliorate psychomotor slowing in schizophrenia over one week?

Participants will complete questionnaires on the first and last day of the study. Each day, participants will receive the TMS-treatment. Optionally, participants can receive a cerebral MRI before the study and/or come for an additional day 6 to repeat some of the questionnaires.

There is no comparison group. All participants will receive the same treatment.

DETAILED DESCRIPTION:
Schizophrenia is a chronic disorder causing tremendous burden to the patients, families, and society. Besides prominent symptoms such as hallucinations, delusions, and thought disorder, the majority of patients also experiences motor abnormalities. Converging evidence links aberrant structure and function of the cerebral motor network to schizophrenia pathology, particularly to motor abnormalities. One of the most frequent motor abnormalities is psychomotor slowing (PS), which may impact both gross and fine motor behaviour. While PS causes significant distress and predicts poor outcome, researchers are just starting to understand its pathobiology. First evidence points to aberrant functional and structural connectivity within the cerebral motor network in schizophrenia patients with PS, particularly in connections between premotor/motor cortex and thalamus, as well as between motor cortex and cerebellum. In addition, severe motor inhibition was linked to increased neural activity in the premotor cortex. Repetitive transcranial magnetic stimulation (rTMS) may temporarily alter brain activity.

Data from OCoPS-P (BASEC 2018-02164, clinicaltrials.gov NCT03921450) double-blind RCT indicate that 15 sessions of inhibitory rTMS over three weeks on the supplementary motor area (SMA) alleviate PS.

However, three weeks of one daily rTMS session is rather inconvenient for patients and medical professionals. Therefore, this study will aim to optimize the treatment protocol with regard to efficiency and efficacy by using an accelerated rTMS protocol with continuous theta-burst stimulation (cTBS). Inhibitory cTBS will be applied 3 times per day over 5 days, which will increase the session frequency and shorten sessions and treatment duration.

Reducing the duration of the treatment phase might increase treatment adherence, shorten inpatient treatment, alleviate PS faster, and will facilitate implementation in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years.
* Ability and willingness to participate in the study
* Ability to provide written informed consent
* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Schizophrenia spectrum disorders according to DSM-5 with psychomotor slowing (SRRS score ≥ 15).

Exclusion Criteria:

* Substance abuse or dependence other than nicotine.
* Past or current medical or neurological conditions associated with impaired or aberrant movement, such as brain tumors, stroke, M. Parkinson, M. Huntington, dystonia.
* Severe head trauma with subsequent loss of consciousness.
* Epilepsy or other convulsions.
* History of any hearing problems or ringing in the ears.
* Standard exclusion criteria for TMS (implanted electronic devices (e.g. pacemakers, implantable cardioverter-defibrillators, vagus nerve stimulators and wearable cardioverter-defibrillators, ocular implants, deep brain stimulators, implanted medication pumps, intracardiac lines even when removed) and/or conductive objects near the coil (e.g. cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents and bullet fragments)
* Women who are pregnant or breastfeeding.
* Any TMS treatment in the past 2 months.
* If applicable: standard exclusion criteria for MRI (study participation without MRI is possible)
* Intention to become pregnant during the course of the study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees, and other dependent persons

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Salpetriere Retardation Rating Scale (SSRS) from baseline | At baseline, day 3, post at day 5, and follow-up 1 week later
  Changes in psychomotor slowing as measured by the Salpêtrière retardation rating scale (SRRS) throughout the study.
  The SRRS is a 15-item rating scale that measures psychomotor slowing. Each item can be scored from 0 to 4, thus the total ranging from 0 to 60, with lower scores representing better outcome.
Proportion of responders in SRRS | At baseline, day 3, post at day 5, and follow-up 1 week later
  Proportion of responders (>= 30% reduction from baseline SRRS) at day 3 and day 5. This will provide an additional categorical measure of who benefits from the intervention in terms of the main target (psychomotor slowing).

SECONDARY OUTCOMES:
Change in psychosis severity from baseline | At baseline, post at day 5, and follow-up 1 week later
  Change in the Positive And Negative Symptom Scale (PANSS) from baseline, PANSS total score assesses the severity of positive, negative and general symptoms, ranging from 30-210 with higher scores indicating increased symptom severity, i.e. poorer outcome
Change in negative symptoms from baseline | At baseline, post at day 5, and follow-up 1 week later
  Change in the Brief Negative Symptom Scale (BNSS) from baseline, total score is used, ranging from 0-78 with higher values indicating poorer outcome, i.e. more negative symptom severity
Change in catatonia severity from baseline | At baseline, day 3, post at day 5, and follow-up 1 week later
  Observer based rating of catatonia severity with the Bush Francis Catatonia Rating Scale (BFCRS), total score of the BFCRS ranging 0-69, with higher scores indicating poorer outcome Observer based rating of catatonia severity with the Northoff Catatonia Rating Scale (NCRS), total score ranging 0-80, with higher scores indicating poorer outcome
Change in parkinsonism severity from baseline | At baseline, day 3, post at day 5, and follow-up 1 week later
  Observer based rating of parkinsonism severity with the Unified Parkinson Disease Rating Scale Part III (UPDRS), total score of the UPDRS ranging 0-104, with higher scores indicating poorer outcome
Changes in neurological soft signs from baseline | At baseline, post at day 5, and follow-up 1 week later
  Observer based rating of neurological soft signs with the Neurological Evaluation Scale (NES), total score ranging 0-82, with higher scores indicating poorer outcome
Changes in dyskinesia from baseline | At baseline, post at day 5
  Observer based rating of dyskinesia with the Abnormal Involuntary Movement Scale (AIMS), 7-item scale with the total ranging fro 0-28, with higher scores indicating poorer outcome
Changes in self-reported negative symptoms from baseline | At baseline, post at day 5
  Self-reported negative symptoms with the Self-evaluation of Negative Symptoms (SNS), total score ranging 0-40, with higher scores indicating poorer outcome
Changes in self-reported catatonia symptoms from baseline | At baseline, post at day 5
  Self-reported catatonia symptoms with the Northoff Scale for Subjective Experience in Catatonia (NSSC), total score ranging 0-48, with higher scores indicating poorer outcome
Changes in self-reported activity from baseline | At baseline, post at day 5
  Change in the International Physical Activity Questionnaire (IPAQ), the total score is used ranging from 0-70000 metabolic equivalent (MET)
Change in objectively measured physical activity from baseline | Continuously from baseline to post at day 5
  Change in the activity levels using wrist actigraphy from baseline. Actigraphy is measured continuously from baseline to post and a sleep diary is collected to separate wake from sleep hours
Change in dexterity from baseline | At baseline, post at day 5
  Change in the coin rotation task from baseline
Change in grip strength from baseline | At baseline, post at day 5
  Change in grip strength measured with a grip force task
Change in cortical excitability of the motor cortex from baseline | Baseline before the first 3 TMS, baseline after the first 3 TMS, day 3 (after 9 TMS), post at day 5 (after 15 TMS)
  Changes in motor cortex excitability from beginning of day 1, end of day 1, end of day 3, and end of day 5 using a TMS paradigm of short interval intracortical inhibition (SICI), intracortical facilitation (ICF) and 1 mV motor evoked potentials (MEP).
Change in social and community functioning | Baseline, post at day 5
  Change in Social and Occupational Functional Assesment Scale (SOFAS) from baseline, the score ranges from 0-100 with higher scores indicating better functioning, i.e. better outcome
Change in global functioning | Baseline, post at day 5
  Change in Global Assessment of Functioning (GAF) from baseline, total score ranging 0-100 with higher scores indicating better functioning/outcome
Change in functional capacity | Baseline, post at day 5
  Change in the Score of the brief version of the University of California, San Diego, Performance-Based Skills Assessment (UPSA-brief) assessment from baseline, higher scores indicating better function, the total score is used ranging 0-100
Change in DSM 5 Severity Scale of Dimensions | Baseline, post at day 5
  Change in expert rated DMS 5 Severity Scale of Dimensions from baseline. Eight symptom dimensions are rated from 0 to 4 (total 0-32), with higher scores indicating worse outcomes

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by a safety questionnaire | Daily between baseline and post at day 5
  After all TMS sessions of one day (after 3, 6, 9, 12, and 15 cTBS sessions) the investigators will apply a short safety questionnaire to assess the incidence of the most common side effects of TMS.
Incidence of spontaneously mentioned Treatment-Emergent Adverse Events | Daily between baseline and post at day 5, and follow-up 1 week later
  After each cTBS session, participants are inquired about stimulation side effects (Adverse Events and Device Deficiencies) with the unspecific question "was anything uncomfortable during the stimulation?".
Resting-state functional connectivity as a Biomarker of the severity of PS | In the week before baseline
  Regression analyses between the clinical assessment of PS severity (assessed by the motor rating scales and the objective measurements) and the resting state functional connectivity (using resting-state BOLD fMRI) within the cerebral motor system
Resting state cerebral perfusion as a Biomarker of the severity of PS | In the week before baseline
  Regression analyses between the clinical assessment of PS severity (assessed by the motor rating scales and the objective measurements) and the resting state cerebral perfusion (using resting-state cerebral perfusion fMRI) within the cerebral motor system
Structural connectivity as a Biomarker of the severity of PS | In the week before baseline
  Regression analyses between the clinical assessment of PS severity (assessed by the motor rating scales and the objective measurements) and the structural integrity of the sensory motor pathway using the diffusion MRI data.
Resting-state functional connectivity as a Biomarker of the response to cTBS | In the week before baseline
  Comparison of the resting state functional connectivity (using resting-state BOLD fMRI) within the cerebral motor system between the patients who responded (evaluated with the % of change in SRRS) or not to cTBS
Resting state cerebral perfusion as a Biomarker of the severity of PS | In the week before baseline
  Comparison of the resting state cerebral perfusion (using resting-state cerebral perfusion fMRI) within the cerebral motor system between the patients who responded (evaluated with the % of change in SRRS) or not to cTBS
Structural connectivity as a Biomarker of the severity of PS | In the week before baseline
  Comparison of the structural integrity of the sensory motor pathway using the diffusion MRI data between the patients who responded (evaluated with the % of change in SRRS) or not to cTBS

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Walther, Prof. Dr. med, Principal Investigator — Translational Research Center, University Hospital of Psychiatry and Psychotherapy, University of Bern, Bern, Switzerland
Locations (1):
- University Hospital of Psychiatry and Psychotherapy, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No